CLINICAL TRIAL: NCT00669474
Title: Unicentric Comparing Study of Suction Curettage With Standard BOTOX Injection in the Treatment of Patients With Essential Axillar Hyperhidrosis: Comparing of Efficacy, Duration of Effectiveness, and Adverse Events.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study never started
Sponsor: University Hospital, Ghent (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008/219
Record Dates: First submitted 2008-04-28; First posted 2008-04-30 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Essential Axillary Hyperhidrosis
MeSH Terms: interventions — Vacuum Curettage; Therapeutics; Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): Suction curettage
  Interventions: Procedure: Suction curettage
- 2 (Active Comparator): Treatment with Botox
  Interventions: Drug: Treatment with Botox

INTERVENTIONS:
Procedure: Suction curettage — Suction curettage
  Arms: 1
Drug: Treatment with Botox — Treatment with Botox
  Arms: 2

SUMMARY:
Part 1: patients with essential hyperhidrosis are treated one time with suction curettage in both axillae.

Part 2: patients with axillary hyperhidrosis receive one treatment with suction curettage in one axilla, and at the same time one treatment with BOTOX injections in the other axilla.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years
* Persistent bilateral primary axillary hyperhidrosis
* Hidrosis interferes with daily activities of patient
* Gravimetrically minimal 50 mg spontaneous sweat production in each axilla, measured during 5 minutes in room temperature in calm condition
* signed informed consent
* patient can and shall continue the trial until the end, and will follow the instructions correcly
* women in reproductive period had a pregnancy test

Exclusion Criteria:

* Medical condition that can be dangerous by treatment with BOTOX, including myastenia gravis, Lambert-Eaton syndrome, ALS, and each other disease that can interfere with the neuromuscular function
* Secundary hyperhidrosis (for example secundary on hyperthyroid problems, lymfoma, malaria)
* Known allergy against study medication, his components, local anesthesia or iodium
* Use of aminoglycosids, curare-like products, or other products which can interfere with the neuromuscular function during the study
* Use of therapy for hyperhidrosis with Aluminium chlorid during the study
* Infection or skin disease in the area to treat
* Participation in an other therapeutic study on the same time
* Botuline toxine treatment in the last 4 months
* Women who can or who want to become pregnant
* Women in reproductive period who don't use the appropriate contraception
* Patients in a situation of which the researchers decide it can be dangerous, or can interfere with the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2009-06; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Effectiviness and duration of effect of both treatments | 1 year

SECONDARY OUTCOMES:
Adverse events of both treatments | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Katia Ongenae, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Related Info — http://www.uzgent.be